CLINICAL TRIAL: NCT04377932
Title: Interleukin-15 Armored Glypican-3-specific Chimeric Antigen Receptor Expressing Autologous T Cells as Immunotherapy for Children With Solid Tumors
Brief Title: Interleukin-15 Armored Glypican 3-specific Chimeric Antigen Receptor Expressed in T Cells for Pediatric Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David Steffin, MD, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H-47757 AGAR
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Liver Cancer; Rhabdomyosarcoma; Malignant Rhabdoid Tumor; Liposarcoma; Wilms Tumor; Yolk Sac Tumor
Keywords: 15.GPC3-CAR T cells; GPC3; Glypican
MeSH Terms: conditions — Liver Neoplasms; Rhabdomyosarcoma; Rhabdoid Tumor; Liposarcoma; Wilms Tumor; Endodermal Sinus Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AGAR T cells (Experimental): GPC3-CAR and the IL15 (AGAR T cells) will be administered to patients with GPC3-positive solid tumors.
  Interventions: Genetic: AGAR T cells

INTERVENTIONS:
Genetic: AGAR T cells — Four different dosing schedules will be evaluated. Three to six patients will be evaluated on each dosing schedule. The following dose levels will be evaluated:
  DL1: 3x10^7/m2 DL2: 1x10^8/m2 DL3: 3x10^8/m2 DL4: 1x10^9/m2
  The doses are calculated according to the actual number of GPC3-CAR transduced T cells.
  Other Names: GPC3-CAR T cells

SUMMARY:
Patients may be considered if the cancer has come back, has not gone away after standard treatment or the patient cannot receive standard treatment. This research study uses special immune system cells called AGAR T cells, a new experimental treatment.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise, but have not been strong enough to cure most patients.

Investigators have found from previous research that they can put a new gene (a tiny part of what makes-up DNA and carries your traits) into T cells that will make them recognize cancer cells and kill them. In the lab, investigators made several genes called a chimeric antigen receptor (CAR), from an antibody called GPC3. The antibody GPC3 recognizes a protein found solid tumors including pediatric liver cancers. This CAR is called GPC3-CAR. To make this CAR more effective, investigators also added a gene that includes IL15. IL15 is a protein that helps CAR T cells grow better and stay in the blood longer so that they may kill tumors better. The mixture of GPC3-CAR and IL15 killed tumor cells better in the laboratory when compared with CAR T cells that did not have IL15 .This study will test T cells that investigators made (called genetic engineering) with GPC3-CAR and the IL15 (AGAR T cells) in patients with GPC3-positive solid tumors such as yours.

T cells made to carry a gene called iCasp9 can be killed when they encounter a specific drug called Rimiducid. The investigators will insert the iCasp9 and IL15 together into the T cells using a virus that has been made for this study. The drug (Rimiducid) is an experimental drug that has been tested in humans with no bad side-effects. The investigators will use this drug to kill the T cells if necessary due to side effects.

This study will test T cells genetically engineered with a GPC3-CAR and IL15 (AGAR T cells) in patients with GPC3-positive solid tumors.

The AGAR T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the biggest dose of AGAR T cells that is safe, to see how long they last in the body, to learn what the side effects are and to see if the AGAR T cells will help people with GPC3-positive solid tumors.

DETAILED DESCRIPTION:
Approximately 15-24 subjects will participate in the treatment part of this study.

Maximum of 180 mL of blood (not exceeding 3ml/kg/day) is collected from patients to grow the T cells and a retrovirus (a special virus that can insert the GPC3 CAR gene into the T cells) is used to genetically engineer them. After the CAR gene was put into the T cells, the investigators make sure that they are able to kill GPC3 positive solid tumor cells in the laboratory.

LYMPHODEPLETION CHEMOTHERAPY:

Several studies suggest that the infused T cells need room to be able to increase in numbers/multiply and accomplish their functions and that this may not happen if there are too many other T cells in circulation . Because of that, participants will receive treatment with lymphodepletion chemotherapy. This chemotherapy means the participant will receive both cyclophosphamide (Cytoxan) and fludarabine. Participants will receive these drugs for 3 days before receiving the T-cell infusion. These drugs will decrease the numbers of the participants own T cells before the investigators infuse the AGAR T cells.

WHAT THE INFUSION WILL BE LIKE:

After making these cells, they will be frozen. If the patient agrees to participate in this study, at the time the patient is scheduled to be treated, the cells will be thawed and injected into the patient over 5 to 10 minutes. The participant will receive the AGAR T CELLS 48 to 72 hours after completing the chemotherapy.

This is a dose escalation study, which means that the investigators do not know the highest dose of GAP T cells that is safe. To find out, the investigators will give the cells to at least 3 participants at one dose level. If that is safe, the investigators will raise the dose given to the next group of participants. The dose each patient gets depends on how many participants get the agent before that patient and how they react. The investigator will tell each patient this information. If your cancer responds to therapy and there are no DLTs, we would allow for up to 3 additional treatments at that same dose. This will help the participant think about possible harms and benefits. Since the treatment is experimental, what is likely to happen at any dose is not known.

All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital.

Medical tests before treatment:

* Physical exam and History
* Blood tests to measure blood cells, kidney and liver function.
* Pregnancy test (if the participant is a female who can get pregnant)
* If the participant is infected with the hepatitis B virus (HBV) the investigators will do a test to measure the levels of the virus
* Measurements of the participant's tumor by scans and the tumor marker alfa-fetoprotein (AFP), if the participant's tumor produces this protein. Tumor markers are molecules in the blood that are higher when a person has certain cancers

Medical tests during and after treatment:

* Physical exams and History
* Blood tests to measure blood cells, kidney and liver function
* If the participant is infected with the hepatitis B virus (HBV) the investigators will repeat the test and monitor the levels of the virus
* Measurements of the participant's tumor by scans (4-6 weeks after the infusion) and AFP (if applicable at 1, 2, and 4 weeks after the infusion).
* Tumor biopsy between 2-4 weeks after the infusion and as clinically indicated thereafter. For additional clinically indicated tumor biopsies, investigators will ask for a portion of the sample for research.

FOLLOW-UP STUDIES The investigators will follow the participant during and after each injection. To learn more about the way the T cells are working in the participant's body, up to 60 mL (upto 12 teaspoons, no more than 3ml/kg/day) of blood will be taken from the participant before the chemotherapy, before the T-cell infusion, 1 to 4 hours after the infusion, 3 to 4 days after the infusion (this time point is optional ) at 1 week, 2 weeks, 4 weeks and 8 weeks after the injection, every 3 months for

1 year, every 6 months for 4 years and then every year for the next 10 years. Total participation time for this study will be 15 years.

During the time points listed above, if the T cells are found in the participant's blood at a certain amount an extra 5 mL of blood may need to be collected for additional testing.

The investigators will use this blood to look for the frequency and activity of the cells that the investigators have given; that is, to learn more about the way the T cells are working and how long they last in the body. The investigators will also use this blood to see if there are any long-term side effects of putting the new gene (chimeric antigen receptor, CAR) into the cells. In addition to the blood draws, because the participants have received cells that have had a new gene put in them, the participants will need to have long term follow up for 15 years so the investigators can see if there are any long-term side effects of the gene transfer.

Once a year, the participants will be asked to have their blood drawn and answer questions about their general health and medical condition. The investigators may ask the participants to report any recent hospitalizations, new medications, or the development of conditions or illness that were not present when the participants enrolled in the study and may request that physical exams and/or laboratory tests be performed if necessary.

When tumor biopsy is performed for clinical reasons the investigators will request permission to obtain excess sample to learn more about the effects of the treatment on the participant's disease.

In the event of death, the investigators will request permission to perform an autopsy to learn more about the effects of the treatment on the participant's disease and if there were any side effects from the cells with the new gene.

In addition, the investigators would like to ask for participant permission to use tumor biopsy for research purposes only. Associated risk with the biopsy will be discussed with each participant in detail in a procedure specific consent form. The investigators will test the sample to see if the GAP T cells can be found in the tumor and what effect they had on the tumor cells.

If participants develop a second abnormal cancer growth, significant blood or nervous system disorder during the trial, a biopsy sample of the tissue will be tested.

ELIGIBILITY:
Procurement Eligibility

Inclusion Criteria:

* Diagnosis of GPC3-positive* solid tumors (as determined by immunohistochemistry with an extent score of >=Grade 2 [>25% positive tumor cells] and an intensity score of >= 2 [scale 0-4]).
* Age ≥ 1 year and ≤ 21 years
* Life expectancy of ≥ 16 weeks
* Lansky or Karnofsky score ≥60%
* Barcelona Clinic Liver Cancer Stage A, B or C (for patients with hepatocellular carcinoma only
* Child-Pugh-Turcotte score <7 (for patients with hepatocellular carcinoma only)
* Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Exclusion Criteria:

* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)
* History of organ transplantation
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* Actively progressing CNS metastases

Treatment Eligibility

Inclusion Criteria:

* Age ≥ 1 year and ≤ 21 years
* Barcelona Clinic Liver Cancer Stage A, B or C (for patients with hepatocellular carcinoma only)
* Lansky or Karnofsky score ≥ 60%
* Child-Pugh-Turcotte score < 7 (for patients with hepatocellular carcinoma only)
* Adequate organ function:
* Creatinine clearance as estimated by Cockcroft Gault or Schwartz ≥ 60 ml/min
* serum AST< 5 times ULN
* total bilirubin < 3 times ULN for age
* INR ≤1.7 (for patients with hepatocellular carcinoma only)
* absolute neutrophil count > 500/microliter
* platelet count > 25,000/microliter (can be transfused but must be at that level prior to treatment)
* Hgb ≥7.0 g/dl (can be transfused but must be at that level prior to treatment)
* pulse oximetry >90% on room air
* Refractory or relapsed disease after treatment with up- front therapy and at least one salvage treatment cycle
* Recovered from acute toxic effects of all prior chemotherapy and investigational agents before entering this study
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 3 months after the T-cell infusion.
* Informed consent explained to, understood by and signed by patient/ guardian. Patient/guardian given copy of informed consent

Exclusion Criteria

* Pregnancy or lactation
* Uncontrolled infection
* Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day, dose adjustment or discontinuation of medication must occur at least 24 hours prior to CAR T cell infusion)
* Known HIV positivity
* Active bacterial, fungal or viral infection (except Hepatitis B or Hepatitis C virus infections)
* History of organ transplantation
* History of hypersensitivity reactions to murine protein-containing products OR presence of human anti-mouse antibody (HAMA) prior to enrollment (only patients who have received prior therapy with murine antibodies)
* Actively progressing CNS metastases

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2040-08-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David Steffin, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 15.GPC3-CAR T Cells - Dose Level 1: Participants with GPC3-positive solid tumors received an intravenous injection of 15.GPC3-CAR T cells at Dose Level 1 (3x10^7/m2) after lymphodepleting chemotherapy. The dose was calculated according to the actual number of GPC3-CAR transduced T cells.
- 15.GPC3-CAR T Cells - Dose Level 2: Participants with GPC3-positive solid tumors received an intravenous injection of 15.GPC3-CAR T cells at Dose Level 2 (DL2: 1x10^8/m2) after lymphodepleting chemotherapy. The dose was calculated according to the actual number of GPC3-CAR transduced T cells.
- 15.GPC3-CAR T Cells - Dose Level 3: Participants with GPC3-positive solid tumors received an intravenous injection of 15.GPC3-CAR T cells at Dose Level 3 (DL3: 3x10^8/m2) after lymphodepleting chemotherapy. The dose was calculated according to the actual number of GPC3-CAR transduced T cells.
Period: Dose Level 1
Arm/Group | 15.GPC3-CAR T Cells - Dose Level 1 | 15.GPC3-CAR T Cells - Dose Level 2 | 15.GPC3-CAR T Cells - Dose Level 3
Started | 8 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 8 | 0 | 0
Not completed — Death | 7 | 0 | 0
Not completed — On long term follow up | 1 | 0 | 0
Period: Dose Level 2
Arm/Group | 15.GPC3-CAR T Cells - Dose Level 1 | 15.GPC3-CAR T Cells - Dose Level 2 | 15.GPC3-CAR T Cells - Dose Level 3
Started | 0 | 3 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 3 | 0
Not completed — Death | 0 | 3 | 0
Period: Dose Level 3
Arm/Group | 15.GPC3-CAR T Cells - Dose Level 1 | 15.GPC3-CAR T Cells - Dose Level 2 | 15.GPC3-CAR T Cells - Dose Level 3
Started | 0 | 0 | 3
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 3
Not completed — Death | 0 | 0 | 2
Not completed — On long term follow up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants with GPC3-positive solid tumors received 15.GPC3-CAR T cells.
Groups:
- Total: Total of all reporting groups
Arm/Group | 15.GPC3-CAR T Cells - Dose Level 1 | 15.GPC3-CAR T Cells - Dose Level 2 | 15.GPC3-CAR T Cells - Dose Level 3 | Total
Number analyzed (Participants) | 8 | 3 | 3 | 14
Age, Continuous [Median (Full Range); unit: years] | 10.5 [6.0 to 20.0] | 4.0 [4.0 to 12.0] | 11.0 [5.0 to 20.0] | 10.5 [4.0 to 20.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 2 | 6
  Male | 4 | 3 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 3 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 6 | 2 | 2 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicity
Description: A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the GPC3-CAR T cells. Specifically those which are Grade 5; non-hematologic Grade 3-4 not returning to Grade 2 within 72 hours; Grade 2-4 allergic reaction; grade 4 hematologic toxicity that persists for 28 days or greater; all grade 4 CRS and neurologic toxicities and grade 3 CRS and neurologic toxicities that fail to return to Grade 1 within 7 days.
Time Frame: 4 weeks
Population: Analysis population included participants who received 15.GPC3-CAR T cells and were evaluable for dose limiting toxicity (DLT), defined as those who developed DLTs or completed the 4-week DLT evaluation period after the T cell infusion. One participant at dose level 3 did not complete the DLT evaluation and was not evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | 15.GPC3-CAR T Cells - Dose Level 1 | 15.GPC3-CAR T Cells - Dose Level 2 | 15.GPC3-CAR T Cells - Dose Level 3
Number analyzed (Participants) | 8 | 3 | 2
Participants | 1 | 0 | 0

2. Secondary Outcome: Response Rate
Description: Response rate is calculated as the percentage of subjects with the best overall response that is either complete response or partial response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 4 weeks
Population: Analysis population included participants who received 15.GPC3-CAR T cells and had available response data . One participant at dose level 3 was excluded because response data were not available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 15.GPC3-CAR T Cells - Dose Level 1 | 15.GPC3-CAR T Cells - Dose Level 2 | 15.GPC3-CAR T Cells - Dose Level 3
Number analyzed (Participants) | 8 | 3 | 2
Percentage of participants | 50.0 [15.7 to 84.3] | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7]

3. Secondary Outcome: Maximum Tolerated Dose (MTD) of Autologous Glypican-3 Specific Chimeric Antigen Expressing T Cells Co-expressing IL-15 Administered to Patients With GPC3-positive Solid Tumors.
Description: Defined as the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate. If there is no DLT that determine a MTD, the maximum dose level will be declared as the MTD. In case the lowest dose level is determined to be too toxic and the elimination boundary is reached, no MTD will be defined for the trial.
Time Frame: 28 days
Population: Analysis population included all participants who received 15.GPC3-CAR T cells and were evaluable for DLT, defined as those who developed DLTs or completed the 4-week DLT evaluation period after the T cell infusion. One participant at dose level 3 was excluded because the participant did not complete the DLT evaluation period and was not evaluable for DLT.
Measure: Number; unit: 10^8 cells per square meter
Groups:
- 15.GPC3-CAR T Cells - All Dose Levels (DLT- Evaluable Population): All participants with GPC3-positive solid tumors received a 15.GPC3-CAR T cell infusion after lymphodepleting chemotherapy and were evaluable for DLT. These participants were monitored across all dose levels, including 8 at Dose Level 1, 3 at Dose Level 2 and 2 at Dose Level 3 (total=13).
  Doses:
  Dose Level 1: 3x10^7/m2 Dose Level 2: 1x10^8/m2 Dose Level 3: 3x10^8/m2
  The doses were calculated according to the actual number of GPC3-CAR transduced T cells.
Arm/Group | 15.GPC3-CAR T Cells - All Dose Levels (DLT- Evaluable Population)
Number analyzed (Participants) | 13
10^8 cells per square meter | 3.0

ADVERSE EVENTS:
Time Frame: Data on adverse experiences/toxicities regardless of seriousness were collected for documentation purposes only for 4 weeks after the last dosing of the study drug/biologic.
Arm/Group | 15.GPC3-CAR T Cells - Dose Level 1 | 15.GPC3-CAR T Cells - Dose Level 2 | 15.GPC3-CAR T Cells - Dose Level 3
All-Cause Mortality (participants affected / at risk) | 7/8 | 3/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 6/8 | 2/3 | 2/3
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15.GPC3-CAR T Cells - Dose Level 1 (N=8) | 15.GPC3-CAR T Cells - Dose Level 2 (N=3) | 15.GPC3-CAR T Cells - Dose Level 3 (N=3)
Ear and labyrinth disorders - Other, specify : phonophobia (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders and administration site conditions) | 5 (8) | 2 (10) | 2 (3)
Flu like symptoms (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 5 (14) | 2 (2) | 2 (3)
Infections and infestations-Other,specify:Bacteremia due to e.coli. without vomiting or diarrhea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify : budding yeast infection at vascular access port (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify : Disease progression to the brain and nervous system (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify : cerebral hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify : neurologic failure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15.GPC3-CAR T Cells - Dose Level 1 (N=8) | 15.GPC3-CAR T Cells - Dose Level 2 (N=3) | 15.GPC3-CAR T Cells - Dose Level 3 (N=3)
Anemia (Blood and lymphatic system disorders) | 7 (10) | 2 (4) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (10) | 3 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (3) | 1 (1)
Chills (General disorders and administration site conditions) | 1 (1) | 2 (3) | 1 (1)
Edema face (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (2)
Edema limbs (General disorders and administration site conditions) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders and administration site conditions) | 3 (4) | 2 (6) | 2 (2)
Fever (General disorders and administration site conditions) | 5 (9) | 1 (8) | 0 (0)
Non-cardiac chest pain (General disorders and administration site conditions) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 1 (2) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (8) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (8) | 2 (2) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3) | 2 (3) | 2 (2)
Creatinine increased (Investigations) | 5 (5) | 1 (2) | 0 (0)
GGT increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
INR increased (Investigations) | 2 (2) | 1 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 8 (11) | 3 (5) | 3 (3)
Neutrophil count decreased (Investigations) | 8 (11) | 3 (5) | 3 (3)
Platelet count decreased (Investigations) | 7 (10) | 3 (5) | 2 (2)
White blood cell decreased (Investigations) | 8 (10) | 3 (5) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (10) | 3 (4) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (7) | 1 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (10) | 2 (3) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 6 (8) | 1 (2) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (6) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 6 (8) | 2 (4) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify : mild chest pain upon inhalation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : Genital Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : HSV+ ulcers in mouth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify : Periorbital Edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT04377932/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT04377932/ICF_001.pdf